CLINICAL TRIAL: NCT00757666
Title: Assessment of Proper Physiologic Response With Rate Adaptive Pacing Driven by Minute Ventilation or Accelerometer
Brief Title: APPROPRIATE - Rate Adaptive Pacing Sensor
Acronym: APPROPRIATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrollment; higher than planned patient attrition and data attrition
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-CA-082808-B
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Heart Diseases
Keywords: Pacemaker
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accelerometer (Active Comparator): Patients implanted with a Boston Scientific ALTRUA 60 pacemaker with accelerometer (motion-based) sensor.
  Interventions: Device: Rate adaptive pacemaker
- Minute Ventilation (Active Comparator): Patients implanted with a Boston Scientific ALTRUA 60 pacemaker with minute ventilation sensor.
  Interventions: Device: Rate adaptive pacemaker

INTERVENTIONS:
Device: Rate adaptive pacemaker — Accelerometer sensor
  Arms: Accelerometer
Device: Rate adaptive pacemaker — Minute ventilation sensor
  Arms: Minute Ventilation

SUMMARY:
The APPROPRIATE study will compare differences in functional capacity (peak VO2) between chronotropically incompetent patients randomized to receive rate responsive pacing driven by either the minute ventilation (respiration-based) sensor or an accelerometer (motion-based).

ELIGIBILITY:
Inclusion Criteria:

* Meets or met current pacemaker implantation indications
* Willing and capable of providing informed consent for participation
* Receiving a dual-chamber pacemaker or previously received a dual-chamber pacemaker with active atrial and ventricular leads
* Plans to remain in the long-term care of his/her enrolling physician and is available for study follow-up for three months post-enrollment

Exclusion Criteria:

* Mobitz II second degree heart block
* Third degree heart block
* Chronic atrial fibrillation or uncontrolled atrial arrhythmias within the past 90 days prior to consent
* Neuromuscular, orthopedic, or vascular disability that prevents normal walking or weight carrying (e.g., intermittent claudication, arthritis, residual stroke weakness, need for a wheelchair or walker)
* A symptom-limited exercise protocol is thought to be dangerous or contra-indicated, including but not limited to changing pattern of chest discomfort or uncontrolled arrhythmias
* Pulmonary disease as defined by any one of the following:

  * Forced Vital Capacity (FVC) or Forced Expiratory Volume in one second (FEV1) < 60% of predicted values
  * Use of two or more pulmonary inhalers
  * Use of supplemental oxygen
  * Chronic use of oral steroids for pulmonary disease treatment
* Life expectancy is less than 12 months due to other medical conditions, per physician discretion
* Has or indicated for an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy-defibrillator (CRT-D)
* Currently enrolled in another investigational study that would directly impact the treatment or outcome of the current study.
* Younger than 18 years of age
* Pregnant or planning to become pregnant during the study (method of assessment upon physician's discretion)
* Unable or unwilling to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Giudici, MD, Principal Investigator — Genesis Heart Institute; F. Roosevelt Gilliam, MD, Principal Investigator — Cardiology Associates of NE Arkansas
Locations (2):
- United States (2):
  - Cardiology Association of NE Arkansas, Jonesboro, Arkansas
  - Genesis Heart Institute, Davenport, Iowa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Accelerometer: Accelerometer
- Minute Ventilation: Minute ventilation
Period: Overall Study
Arm/Group | Accelerometer | Minute Ventilation
Started (566 subjects enrolled, of which 68 had all visits completed at the time of study termination.) | 34 | 34
Completed | 12 (Number of patients with complete CPX test results from 1 month and 2 month visits) | 11 (Number of patients with complete CPX test results from 1 month and 2 month visits)
Not Completed | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Accelerometer | Minute Ventilation | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (8.4) | 70.7 (8.2) | 70.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 21 | 18 | 39
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 68

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Functional Capacity (Peak VO2).
Description: The APPROPRIATE Study compared differences in functional capacity (peak VO2) between CI patients randomized to receive rate responsive pacing driven by either the minute ventilation (respiration-based) sensor or by an accelerometer (motion-based) sensor.
  The mean change in functional capactity will be compared against baseline; changes from baseline will be measured.
Time Frame: 1 month and 2 months post-implant
Population: Data was not analyzed since patient enrollment was ceased and study was prematurely terminated.
Arm/Group | Minute Ventilation | Accelerometer
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Changes in Heart Rate During Activities of Daily Living (ADL) Using a Lift and Carry Test
Description: This outcome measure will be compared against baseline.
Time Frame: 2 months post-implant
Population: Data was not analyzed since patient enrollment was ceased and study was prematurely terminated.
Arm/Group | Accelerometer | Minute Ventilation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Metabolic Chronotropic Relationship (MCR) Slope
Time Frame: 1 month and 2 months post-implant
Population: Data was not analyzed since patient enrollment was ceased and study was prematurely terminated.
Arm/Group | Accelerometer | Minute Ventilation
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

4. Secondary Outcome: Exercise Time
Time Frame: 1 month and 2 months post-implant
Population: Data was not analyzed since patient enrollment was ceased and study was prematurely terminated.
Arm/Group | Accelerometer | Minute Ventilation
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

5. Secondary Outcome: VO2 at Ventilatory Threshold
Time Frame: 1 month and 2 months post-implant
Population: Data was not analyzed since patient enrollment was ceased and study was prematurely terminated.
Arm/Group | Accelerometer | Minute Ventilation
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Accelerometer | Minute Ventilation
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 6/34 | 8/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Accelerometer (N=34) | Minute Ventilation (N=34)
Cardiovascular Adverse Events (Cardiac disorders) | 6 | 8

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. As the study was stopped early, the primary objective is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the results shall be made a joint, multi-center publication.